CLINICAL TRIAL: NCT01191021
Title: Pilot Study to Estimate Central Propofol Effect by Measuring Exhaled Propofol Concentrations
Brief Title: Monitoring Exhaled Propofol to Individualize General Anesthesia
Acronym: EPIGA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: H54427-35579
Record Dates: First submitted 2010-07-20; First posted 2010-08-30 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: General Anesthesia
Keywords: breath; propofol; general anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Propofol (Other): Volunteers will receive propofol anesthesia on the study day.
  Interventions: Drug: Propofol Anesthesia

INTERVENTIONS:
Drug: Propofol Anesthesia — Volunteers will undergo propofol anesthesia for 90 min.

SUMMARY:
This trial investigates the relationship between concentrations of the anesthetic drug propofol in exhaled breath, blood and drug effect in volunteers undergoing general anesthesia. The main goal of this study is to develop a pharmacokinetic - and dynamic model for propofol in exhaled breath.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age

  * Written informed consent
  * Ability and willingness to give written informed consent
  * American Society of Anesthesiologists (ASA) risk score I

Exclusion Criteria:

* Volunteers ASA physical status II - III
* Pregnancy
* Volunteers with history of neurological disease or stroke
* Volunteers with a history of recreational drug abuse
* Volunteers with a history of alcohol abuse
* Smokers
* Anesthesia within 6 months
* Known drug allergies
* History of adverse events during general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Exhaled propofol (parts per billion) | Continuous measurement over 90 min
Processed electroencephalography (Bispectral Index (0-100)): Change from baseline during anesthesia | continuous over 90 min

CONTACTS AND LOCATIONS:
Overall Officials: Christian C Apfel, MD, PhD, Principal Investigator — Perioperative Clinical Research Core, Department of Anesthesia, University of California San Francisco; Cyrill Hornuss, MD, Principal Investigator — Perioperative Clinical Research Core, Department of Anesthesia, University of California San Francisco
Locations (1):
- Department of Anesthesia and Perioperative Care, UCSF, San Francisco, California, United States

REFERENCES:
- [Background] Hornuss C, Praun S, Villinger J, Dornauer A, Moehnle P, Dolch M, Weninger E, Chouker A, Feil C, Briegel J, Thiel M, Schelling G. Real-time monitoring of propofol in expired air in humans undergoing total intravenous anesthesia. Anesthesiology. 2007 Apr;106(4):665-74. doi: 10.1097/01.anes.0000264746.01393.e0. PMID 17413903